CLINICAL TRIAL: NCT06205719
Title: Effect of Remazolam on Anesthesia Recovery in Patients Undergoing Fundus Surgery-A Single-center, Prospective, Randomized, Double-blind, Controlled Clinical Trial
Brief Title: Effect of Remazolam on Anesthesia Recovery in Patients Undergoing Fundus Surgery
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Ting Xu, Principal Investigator, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2023-234-1
Record Dates: First submitted 2024-01-02; First posted 2024-01-16 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Remazolam Anesthesia; Postoperative Recovery
MeSH Terms: interventions — (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol; Flumazenil; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Remazolam combined with Remifentanil anesthesia (Experimental): 0.2mg/kg Remazolam and 2ug/kg Remifentanil for induction of anesthesia, remifentanil 0.1 μg/kg/min and 0.2mg/kg Remazolam were continuously pumped intravenously.
  Interventions: Drug: Remazolam; Drug: Remifentanil
- ciprofol combined with Remifentanil anesthesia (Active Comparator): 0.4mg/kg ciprpfol and 2ug/kg Remifentanil for induction of anesthesia,remifentanil 0.1 μg/kg/min and 0.4-2.4mg/kg/h ciprpfol were continuously pumped intravenously.
  Interventions: Drug: ciprofol; Drug: Remifentanil
- The flumazenil was injected at the end of the surgery (Active Comparator): 0.2mg/kg Remazolam and 2ug/kg Remifentanil for induction of anesthesia, remifentanil 0.1 μg/kg/min and 0.2mg/kg Remazolam were continuously pumped intravenously. The 0.5mg flumazenil was injected at the end of the surgery
  Interventions: Drug: Remazolam; Drug: Flumazenil; Drug: Remifentanil

INTERVENTIONS:
Drug: ciprofol — sedation
  Other Names: haisco pharmaceutical group
  Arms: ciprofol combined with Remifentanil anesthesia
Drug: Remazolam — sedation
  Other Names: Yichang Humanwell Pharmaceutical Company
  Arms: Remazolam combined with Remifentanil anesthesia; The flumazenil was injected at the end of the surgery
Drug: Flumazenil — antagonism
  Other Names: Enwa Pharmaceutical Company
  Arms: The flumazenil was injected at the end of the surgery
Drug: Remifentanil — 2ug/kg Remifentanil
  Other Names: Yichang Humanwell Yichang Humanwell Pharmaceutical Company

SUMMARY:
to investigate the effect of remazolam benzenesulfonate in patients with ocular fundus surgery, so as to guide clinical anesthesiologists to choose more appropriate anesthetic drugs in fundus surgery

DETAILED DESCRIPTION:
to investigate the effect of remazolam benzenesulfonate in patients with ocular fundus surgery, so as to guide clinical anesthesiologists to choose more appropriate anesthetic drugs in fundus surgery。There are three groups.In Group H, ciprofol + Remifentanil was used for maintenance of anesthesia, in Group R, remifentanil + Remifentanil was used for maintenance of anesthesia, in Group RF, remifentanil + Remifentanil was used for maintenance of anesthesia, at the end of the operation, flumazenil was used to counteract the residual anesthetic effect.The quality of postoperative recovery was compared

ELIGIBILITY:
Inclusion Criteria:

1. ASA I-II, patients
2. aged 18-65 years old;
3. Fundus surgery to be performed under general anesthesia ;
4. The expected duration of surgery is about 30-120 min ;
5. BMI: 18-30 kg/m2 ;
6. Those who signed the informed consent form and volunteered to participate in this trial

Exclusion Criteria:

1. Patients with known or suspected genetic susceptibility to malignant hyperthermia;
2. Patients with history of asthma;
3. Patients with severe heart diseases (NYHA ≥ III, severe arrhythmia, etc.) and cerebral or pulmonary diseases, liver or kidney dysfunction; or with unstable vital signs;
4. Patients with history of long-term narcotic analgesics application, including sedative and antidepressant drugs;
5. Patients with history of psychotropic drug abuse within 3 months;
6. Patients with long-term alcohol abuse;
7. People with mental disorder and unable to communicate normally;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
time for recovery | 3 second to 30minutes
  The time from stopping the anesthetic to waking up

CONTACTS AND LOCATIONS:
Overall Officials: Ting Xu, Principal Investigator — Sichuan provincial Peopel'Hospital